CLINICAL TRIAL: NCT01124097
Title: A Phase 3, Double Blind, Randomized, Placebo Controlled, Parallel Group, Multicenter Clinical Study of Eslicarbazepine Acetate in Post-Herpetic Neuralgia
Brief Title: Eslicarbazepine Acetate as Therapy in Post-Herpetic Neuralgia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-308; 2010-019101-42 (EudraCT Number)
Record Dates: First submitted 2010-05-03; First posted 2010-05-14 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Post Herpetic Neuralgia
Keywords: post herpetic neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eslicarbazepine acetate 800 mg once daily (QD) (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Eslicarbazepine acetate 1200 mg QD (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Eslicarbazepine acetate 1600 mg QD (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate (BIA 2-093) — Tablets will be used.
  Other Names: Exalief; Zebinix; BIA 2-093; ESL
  Arms: Eslicarbazepine acetate 1200 mg QD; Eslicarbazepine acetate 1600 mg QD; Eslicarbazepine acetate 800 mg once daily (QD)
Drug: Placebo — Tablets will be used.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of Eslicarbazepine acetate (ESL) as therapy in subjects with Post-herpetic Neuralgia (PHN) over a 15 week treatment phase.

DETAILED DESCRIPTION:
Post-herpetic neuralgia (PHN) is a syndrome of intractable pain following an acute infection of herpes zoster (shingles).

Treatment for PHN is often suboptimal. More than 50% of the subjects fail to respond to pharmacological treatments or experience intolerable side effects.

The clinical development of ESL to treat neuropathic pain is based on its chemical and pharmacodynamic relationship to sodium channel blockers, including carbamazepine, which is effective for treating some neuropathic pain conditions. Preclinical data supports the theoretical background.

This study will examine the efficacy, safety, tolerability and pharmacokinetics of Eslicarbazepine acetate for the treatment of post herpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 18 years or older. Female subjects are of nonchildbearing potential, defined as surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or at least 2 years postmenopausal (spontaneous amenorrhea for at least 24 months before Visit 1), or if of childbearing potential, subjects agree to use a medically acceptable nonhormonal method of contraception.
* Experiencing pain for at least 6 months after the healing of a herpes zoster skin rash.
* A mean score between 4.0 and 9.0, inclusive, on the 24 hour average pain intensity assessment.
* Compliance with patient diary completion.
* If not used to treat PHN, subjects are permitted to take nonsteroidal anti inflammatory drugs and selective serotonin reuptake inhibitors if they were kept on a stable dose for 1 month prior to Screening and are foreseen to remain stable throughout the study.
* Competent and able to freely give own informed consent.
* Female subjects of childbearing potential, who are not currently breastfeeding, must have a negative serum pregnancy test at Visit 1.

Exclusion Criteria:

* Historical exposure to drugs known to cause neuropathy
* Significant skin lesions (active infection, ulcer, etc).
* Known intolerance to ESL or to other carboxamide derivatives (eg, carbamazepine or oxcarbazepine) or frequent or severe allergic reactions with multiple medications.
* Subjects who previously participated in a clinical study with ESL.
* Major psychiatric disorder.
* Serious or unstable cardiovascular disease that could compromise participation or cause hospitalization during the study.
* Second or third degree atrioventricular blockade not corrected with a pacemaker or any clinically significant abnormality in the 12 lead electrocardiogram as determined by the investigator.
* Subjects taking the following drug classes and individual drugs are excluded: benzodiazepines (except short half life sleep agents), skeletal muscle relaxants, orally administered steroids, capsaicin, mexiletine, centrally acting analgesics (dextromethorphan, tramadol), opiates, topical lidocaine, anticonvulsants, tricyclic antidepressants, and serotonin norepinephrine reuptake inhibitors. These drugs require a minimum washout period of at least 5 times the half life and should be tapered appropriately using product label instructions as a guide.
* Relevant clinical laboratory abnormality that, in the investigator's opinion, can compromise the subject's safety.
* History of drug abuse or dependence (drug categories defined by DSM IV) within the past year, excluding nicotine and caffeine.
* Subjects who, in the previous 30 days, received treatment with a drug that had not received regulatory approval for any indication at the time of study entry.
* History of recurrent epileptic seizures except febrile seizures.
* History of severe gastroparesis or gastric bypass surgery.
* Neurolytic or neurosurgical treatment for PHN.
* Injected anesthetics or steroid use within 30 days of Visit 1.
* Malignancy within past 2 years.
* History of chronic hepatitis B or C within the past 3 months or human immunodeficiency virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Synexus ClinPharm GmbH, Berlin, State of Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty nine (89) clinical sites in 12 countries
  Study period:
  Date of first admission: 2010.09.28 Date of last visit: 2012.04.23
Groups:
- Esl 1600 mg QD; Esl 1200 mg QD; Esl 800 mg Once Daily (QD): Eslicarbazepine acetate (Esl) (BIA 2-093): Tablets will be used.
Period: Overall Study
Arm/Group | Esl 1600 mg QD | Esl 1200 mg QD | Esl 800 mg Once Daily (QD) | Placebo
Started | 60 | 60 | 60 | 60
Safety Population | 60 | 60 | 60 | 60
Efficacy Population | 52 | 53 | 53 | 51
Completed | 26 | 38 | 40 | 46
Not Completed | 34 | 22 | 20 | 14
Not completed — Withdrawal by Subject | 4 | 3 | 2 | 3
Not completed — Lack of Efficacy | 2 | 3 | 1 | 3
Not completed — Adverse Event | 24 | 15 | 15 | 7
Not completed — Protocol Violation | 2 | 0 | 2 | 1
Not completed — Physician Decision | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esl 1600 mg QD | Esl 1200 mg QD | Esl 800 mg Once Daily (QD) | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (16.71) | 65.4 (14.47) | 65.9 (15.6) | 65.4 (14.43) | 64.9 (15.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 35 | 25 | 107
  Male | 36 | 37 | 25 | 35 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Mean Pain
Description: The efficacy analysis was restricted to the primary efficacy variable in the analysis population. The intended treatment period, starting on the day of the randomization and ending at the efficacy cut-off date (October 31, 2011), was the basis for the analysis.
  The primary efficacy variable was the difference between the mean values of 7 daily pain scores preceding the efficacy cut-off date (endpoint mean pain score), and before randomization (baseline mean pain score), respectively. The daily pain scores were based on the morning response to the 11-point Numeric Rating Pain Scale (NRPS) question relating to average pain intensity over the last 24 hours. The NPRS is an 11-point scale from 0-10 ["0" = no pain; "10" = the most intense pain imaginable]
Time Frame: baseline to endpoint
Population: efficacy population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Esl 1600 mg QD | Esl 1200 mg QD | Esl 800 mg Once Daily (QD) | Placebo
Number analyzed (Participants) | 52 | 53 | 53 | 51
units on a scale | -1.19 (0.290) | -1.34 (0.277) | -0.94 (0.281) | -0.77 (0.293)
Statistical Analysis 1: Comparison: Esl 800 mg Once Daily (QD) vs Placebo; Test type: Superiority or Other; p = 0.9321, Dunnett's test
Statistical Analysis 2: Comparison: Esl 1200 mg QD vs Placebo; Test type: Superiority or Other; p = 0.2610, Dunnett's test
Statistical Analysis 3: Comparison: Esl 1600 mg QD vs Placebo; Test type: Superiority or Other; p = 0.4764, Dunnett's test

ADVERSE EVENTS:
Time Frame: participants were followed an average of 55 weeks (19 weeks DB + 36 weeks OL)
Arm/Group | Esl 1600 mg QD | Esl 1200 mg QD | Esl 800 mg Once Daily (QD) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/60 | 6/60 | 4/60 | 2/60
Other Adverse Events (participants affected / at risk) | 46/60 | 45/60 | 40/60 | 6/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esl 1600 mg QD (N=60) | Esl 1200 mg QD (N=60) | Esl 800 mg Once Daily (QD) (N=60) | Placebo (N=60)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esl 1600 mg QD (N=60) | Esl 1200 mg QD (N=60) | Esl 800 mg Once Daily (QD) (N=60) | Placebo (N=60)
Dizziness (Nervous system disorders) | 13 (15) | 6 (6) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 3 (3) | 11 (11) | 0 (0)
Headache (Nervous system disorders) | 10 (11) | 7 (8) | 3 (4) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7) | 4 (4) | 4 (4) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 3 (4) | 2 (2) | 1 (1)
Fatigue (General disorders) | 6 (6) | 2 (2) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 5 (5) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 2 (4) | 1 (1)
Somnolence (Nervous system disorders) | 3 (4) | 3 (4) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other